CLINICAL TRIAL: NCT00003557
Title: A Phase II Trial of Dolastatin-10 (NSC 376128) Administered as an IV Bolus Every 3 Weeks in Patients With Hepatobiliary Cancer
Brief Title: Dolastatin 10 in Treating Patients With Metastatic Or Recurrent Liver, Bile Duct, or Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9409; UCCRC-9409; NCI-T98-0010
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: advanced adult primary liver cancer; recurrent adult primary liver cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; adult primary hepatocellular carcinoma; cholangiocarcinoma of the gallbladder
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — dolastatin 10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Dolastatin-10 (400 mcg/m2 IV every 3 weeks)
  Interventions: Drug: dolastatin 10

INTERVENTIONS:
Drug: dolastatin 10

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of dolastatin 10 in treating patients with metastatic or recurrent liver, bile duct, or gallbladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate, time to progression, and survival of patients with previously untreated advanced hepatobiliary cancer treated with dolastatin 10. II. Determine the toxicity of this regimen in this patient population.

OUTLINE: This is an open label, multicenter study. Patients receive dolastatin 10 IV bolus every 3 weeks. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression. Patients are followed until death.

PROJECTED ACCRUAL: A total of 14-35 evaluable patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic, locally advanced, or recurrent cancer of the liver (hepatoma), bile duct, or gallbladder (cholangiocarcinoma) Bidimensionally measurable disease The following are not considered measurable lesions: Lesions seen on colonoscopic examination or barium studies Bone metastases CNS lesions CEA, CA19-9, or AFP levels Ascites No CNS disease only No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 OR Platelet count at least 75,000/mm3 in patients with clinically documented sequestration or hemodilution unrelated to primary bone marrow insufficiency Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No significant underlying medical or psychiatric illness No active infections No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer and carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for advanced or metastatic hepatobiliary cancer No other concurrent chemotherapy No concurrent investigational antineoplastic drugs Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to only site of measurable disease At least 6 weeks since prior radiotherapy and recovered No concurrent radiotherapy to any lesion Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1999-01; Primary Completion 2000-06 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (11):
- United States (11):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Illinois Oncology Research Association, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - University of Texas - MD Anderson Cancer Center, Houston, Texas